CLINICAL TRIAL: NCT05235841
Title: Effect of Acupressure on Blood Pressure, Heart Rate and Pain Severity of Patients Underwent Coronary Angiography: A Randomized Controlled Trial
Brief Title: Effect of Acupressure on Blood Pressure, Heart Rate and Pain Severity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Emine Derya Ister, doctoral lecturer, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KahramanmarasSIU2021
Record Dates: First submitted 2021-12-20; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Acute Pain; Blood Pressure
Keywords: Acupressure; Coronary Angiography
MeSH Terms: conditions — Acute Pain | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Randomized two arm (intervention and usual care) clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AG (Experimental): The group that met the criteria of the study and applied acupressure protocol before Coronary Angiography
  Interventions: Other: acupressure
- CG (No Intervention): BEFORE CORONARY ANGIOGRAPHY, THE GROUP WITHOUT ANY INTERVENTION, CONTROL GROUP

INTERVENTIONS:
Other: acupressure — Acupressure is a complementary and supportive approach used in symptom management.
  Arms: AG

SUMMARY:
Objective: The aim of this study was to evaluate the effect of acupressure applied before CA procedure on systolic and diastolic blood pressure, mean arterial pressure, pulse and pain intensity parameters after CA.

Design: The study is a randomized controlled trial. Setting: The study occurred at Cardiology Service (CS) of a Training and Research Hospital in Turkey.

Participants: One hundred patients whomet the research criteria.

DETAILED DESCRIPTION:
Heart disease is the most important cause of mortality and morbidity in developed and developing countries, despite all preventive and therapeutic initiatives and newly developed methods.Besides the drug treatments, interventional procedures are also used to diagnose and treat some heart diseases, which are life-saving and have few risks. CA, one of the interventional methods commonly used for this purpose, is the process of obtaining cine-angiographic images by injecting contrast agents into femoral, brachial, radial, axillary arteries.

People experience fear of death and consequent anxiety because CA is an invasive diagnostic method. There is a lot of uncertainty about the procedure, and the usage of this method in the diagnosis of an organ with high vital importance, such as the heart, causes fear.High levels of stress cause cardiac irritability and increased blood pressure; while anxiety and stress persist, temporary myocardial ischemia, increased heart rate, palpitations, and chest pain may develop.

The aim of nursing care in CA patients is to ensure the relief and comfort of the patient before, during, and after the procedure, to determine and prevent complications that may develop at an early stage.It is noted that reducing anxiety and pain before and after CA is essential in ensuring the stability of vital signs. Acupressure used for this purpose is a non-pharmacological nursing initiative that can relieve and reduce pain and regulate anxiety-related blood pressure. This study evaluates the impact of acupressure applied before CA on systolic and diastolic blood pressure, mean arterial pressure, pulse, and pain severity parameters after CA.

Design: The study was a randomized controlled trial. Setting: The study occurred at Cardiology Service (CS) of a Training and Research Hospital in Turkey.

Participants: One hundred patients, met the research criteria were divided into 50 in the intervention (IG) and 50 in the control group (CG) by simple randomization method.

Intervention: The IG received acupressure and the CG received no acupressure. Acupressure was applied to patients in the IG 30-60 minutes before CA. In the study the Li4, HT7, and Extra 1 acupressure points and repeated measures were selected; pain intensity, systolic and diastolic blood pressure and pulse parameters of the patients were measured three times.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years of age and older
* undergoing the coronary angiography process for the first time
* planned coronary angiography
* be able to communicate

Exclusion Criteria:

* having psychological or mental disorders
* having a limb amputation
* receiveing therapy such as massage or acupressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) (T1) | Baseline
  The patient marks his or her own pain on a 10 cm ruler, with painlessness on one end and the most severe pain on the other.
Visual Analog Scale (VAS) (T2) | 5-15 minutes after coronary angiography
  The patient marks his or her own pain on a 10 cm ruler, with painlessness on one end and the most severe pain on the other.
Visual Analog Scale (VAS) (T3) | 1 hour after the 2nd time VAS assessment
  The patient marks his or her own pain on a 10 cm ruler, with painlessness on one end and the most severe pain on the other.
Blood Pressure (T1) | Baseline
  Digital and Calibrated Blood pressure monitor
Blood Pressure (T2) | 5-15 minutes after coronary angiography
  The pressure exerted by the circulating blood on the vessel wall is called blood pressure.Digital and Calibrated Blood pressure monitor
Blood Pressure (T3) | 1 hour after the 2nd time blood pressure measurement
  The pressure exerted by the circulating blood on the vessel wall is called blood pressure.Digital and Calibrated Blood pressure monitor
Heart Rate (T1) | Baseline
  The pressure exerted by the circulating blood on the vessel wall is called blood.A calibrated pulse-oximeter was used to measure the pulse.
Heart Rate (T2) | 5-15 minutes after coronary angiography
  The pressure exerted by the circulating blood on the vessel wall is called blood.A calibrated pulse-oximeter was used to measure the pulse.
Heart Rate (T3) | 1 hour after the 2nd time heart rate measurement
  The pressure exerted by the circulating blood on the vessel wall is called blood.A calibrated pulse-oximeter was used to measure the pulse.

CONTACTS AND LOCATIONS:
Overall Officials: emine derya ister, pHD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derya Ister E, Altinbas Y. Effect of Acupressure on the Blood Pressure, Heart Rate, and Pain Severity of Patients who Underwent Coronary Angiography: A Randomized Controlled Trial. Altern Ther Health Med. 2023 Oct;29(7):216-221. PMID 36112790